CLINICAL TRIAL: NCT01467713
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Once a Day, TAK-375SL as an Adjunctive Therapy to Treatment-as-Usual in the Maintenance Treatment of Bipolar I Disorder in Adult Patients
Brief Title: Efficacy and Safety of Ramelteon Sublingual as Adjunctive Therapy for Maintenance Treatment of Bipolar I Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision; No Safety Concerns.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-375SL_203; U1111-1124-4675 (Registry Identifier: WHO)
Record Dates: First submitted 2011-11-04; First posted 2011-11-09 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Bipolar Disorder
Keywords: Drug Therapy
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Ramelteon SL placebo-matching, tablets, sublingual (SL) [dissolved under the tongue], once daily, every night at bedtime for up to 9 months.
  Interventions: Drug: Placebo
- Ramelteon SL 0.1 mg (Experimental): Ramelteon SL 0.1 mg, tablets, sublingual, once daily, every night at bedtime for up to 9 months.
  Interventions: Drug: Ramelteon SL
- Ramelteon SL 0.4 mg (Experimental): Ramelteon SL 0.4 mg, tablets, sublingual, once daily, every night at bedtime for up to 9 months.
  Interventions: Drug: Ramelteon SL
- Ramelteon SL 0.8 mg (Experimental): Ramelteon SL 0.8 mg, tablets, sublingual, once daily, every night at bedtime for up to 9 months.
  Interventions: Drug: Ramelteon SL

INTERVENTIONS:
Drug: Ramelteon SL — Ramelteon sublingual (SL) tablets
  Other Names: TAK-375SL
  Arms: Ramelteon SL 0.1 mg; Ramelteon SL 0.4 mg; Ramelteon SL 0.8 mg
Drug: Placebo — Ramelteon sublingual (SL) placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of ramelteon, once nightly before bedtime (QHS), sublingual (SL), in the maintenance treatment of Bipolar I Disorder in adult patients.

DETAILED DESCRIPTION:
TAK-375SL (ramelteon sublingual formulation) is being developed by Takeda Pharmaceutical Company Limited as an adjunctive treatment in the maintenance therapy of bipolar I disorder.

Participants will be seen twice a month for the first two months and then once every month up to the end of the 9-month treatment period. Participants who complete the 9-month treatment period will have a follow-up visit approximately seven days after the last visit. A safety followup phone call will be made 30 days after completion of the 9-month treatment period.

Based on the recommendation of the Independent Data Monitoring Committee which determined that the study data had met pre-determined criteria for futility, Takeda has made a decision to terminate the study. No safety concerns were identified by the Independent Data Monitoring Committee

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant suffers from bipolar I disorder, according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria and is confirmed by the Structured Clinical Interview for DSM Disorders (SCID).
4. The participant is a man or woman aged between 18 and 75 years, inclusive.
5. The participant has an identified caregiver or person responsible (e.g. family member, spouse, case worker or nurse at a residential living (facility) that is considered reliable by the investigator.
6. The most recent mood episode (depression, mania, mixed episode) is within the past 9 months from screening.
7. The participant has been in remission in the opinion of the principal investigator (PI) for at least 8 weeks prior to baseline from their most recent mood episode.
8. The participant has a Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≤12 at the Screening and Baseline visits.
9. The participant has a Young Mania Rating Scale (YMRS) score of ≤10 both at the Screening and Baseline visits.
10. The participant has a Clinical Global Impression Scale - Severity (CGI-S) score of ≤2 at the Screening and Baseline visits.
11. Hamilton Rating Scale for Anxiety (HAM-A) score is ≤21 at Screening and Baseline visits.
12. The participant's medications for bipolar I disorder are stable i.e., no dose adjustment has been made for at least 8 weeks prior to the randomization
13. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent through the duration of the study and for 30 days after the last dose.
14. A female participant of childbearing potential who is sexually active with a non sterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose.

Exclusion Criteria:

1. The participant has received any investigational compound <30 days before Screening or 5 half-lives prior to Screening.
2. The participant has ever received ramelteon in a previous clinical study or has ever used ramelteon.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. The participant has one or more of the following:

   * Any current psychiatric disorder which is the primary focus of treatment other than bipolar I disorder as defined in the DSM-IV-TR, as assessed by the SCID.
   * Current or history of: schizophrenia or any other psychotic disorder, including major depression with psychotic features, bipolar depression with psychotic features (with the exception of psychosis associated with a manic or mixed episode), obsessive-compulsive disorder (OCD), mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
   * Current diagnosis or history of alcohol or other substance abuse (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in full and sustained remission for at three months from the day of screening (Participant must also have negative urine drug screen at Screening and Baseline; only exception is for benzodiazepines and opiates provided the participant has a valid prescription).
   * Current diagnosis or history of alcohol or other substance dependence (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in full and sustained remission for at six months from the day of screening.(Participant must also have negative urine drug screen at Screening and Baseline; only exception is for benzodiazepines and opiates provided the participant has a valid prescription).
   * Presence or history of a clinically significant neurological disorder (including epilepsy) as determined by the investigator.
   * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
   * Any Axis II disorder that might compromise the study.
   * History of Rapid Cycling bipolar disorder: Patients who have more than 8 episodes of mood disorder per year.
5. The participant experienced the first episode of mood disorder after the age of 65 years.
6. The participant is on any other medications other than antidepressants (except fluvoxamine), mood stabilizers (lithium, valproate, lamotrigine), or atypical antipsychotics (risperidone, lithium and/or valproate, the levels should be in the specified range: lithium (serum levels up to 1.2 mEq/L); valproate (serum levels up to 125 mcg/ml) at screening.
7. The participant has received electroconvulsive therapy, vagal nerve stimulation, or repetitive transcranial magnetic stimulation within 6 months prior to Screening.
8. The participant has started receiving formal cognitive or behavioral therapy, systematic psychotherapy within 30 days from screening or plans to initiate such therapy during the study (supportive therapy, marital therapy and bereavement counseling are allowed).
9. The participant has a significant risk of suicide according to the investigator's clinical judgment or has a score ≥5 on item 10 (suicidal thoughts) of the MADRS or has made a suicide attempt in the previous 6 months.
10. The participant is required to take excluded medications or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study.
11. The participant has a clinically significant unstable illness, for example hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, hematological, infectious, dermatological disorder or metabolic disturbance.
12. The participant has a history or current diagnosis of Fibromyalgia, Chronic Fatigue Syndrome, Chronic Pain Syndrome and Sleep apnea.
13. The participant has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication. This criterion does not include those participants with basal cell or stage I squamous cell carcinoma of the skin.
14. The participant has 1 or more laboratory value outside the normal range, based on the blood or urine samples taken at the Screening Visit, that are considered by the investigator to be clinically significant; or the participant has any of the following values at the Screening Visit:

    * A serum creatinine value >1.5 times the upper limits of normal (xULN).
    * A serum total bilirubin value >1.5 xULN.
    * A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2 xULN.
15. The participant has glycosylated hemoglobin (HbA1C) ≥7% at screening and no prior diagnosis of diabetes and/or treatment for diabetes. NOTE: Participants with known diabetes are not excluded.
16. The participant has a thyroid stimulating hormone (TSH) value outside the normal range at the Screening Visit that is deemed clinically significant by the investigator. NOTE: T4 will be checked if TSH is out of range. If T4 is abnormal the participant will be excluded.
17. The participant has clinically significant abnormal vital signs as determined by the investigator.
18. The participant has an abnormal electrocardiogram as determined by the central reader and confirmed as clinically significant by the investigator.
19. The participant has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
20. The participant has a positive urine drug screen. NOTE: Positive urine drug screens for benzodiazepines and opiates for which the participant has a valid prescription will be allowed.
21. The participant has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
22. The participant has a positive urine drug screen. NOTE: Positive urine drug screens for benzodiazepines and opiates for which the participant has a valid prescription will be allowed.
23. The participant, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (155):
- United States (137):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Muscle Shoals, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Bellflower, California
  - Costa Mesa, California
  - Garden Grove, California
  - Harbor City, California
  - Huntington Park, California
  - Irvine, California
  - Lomita, California
  - Long Beach, California
  - Los Angeles, California
  - Murrieta, California
  - National City, California
  - Oceanside, California
  - Orange, California
  - Paramount, California
  - Rancho Cucamonga, California
  - Redondo Beach, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - San Jose, California
  - San Ramon, California
  - Sherman Oaks, California
  - Torrance, California
  - Wildomar, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Coral Gables, Florida
  - Coral Springs, Florida
  - Edgewater, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Miami Lakes, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Port Charlotte, Florida
  - Saint Cloud, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Dunwoody, Georgia
  - East Point, Georgia
  - Smyrna, Georgia
  - Suwanee, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Gurnee, Illinois
  - Libertyville, Illinois
  - Skokie, Illinois
  - Brownsburg, Indiana
  - Manhattan, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Bloomfield Hills, Michigan
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Flowood, Mississippi
  - Hazelwood, Missouri
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Cherry Hill, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Cedarhurst, New York
  - Fresh Meadows, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Columbiana, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Franklin, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - McMurray, Pennsylvania
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Lincoln, Rhode Island
  - Columbia, South Carolina
  - Greer, South Carolina
  - Old Point Station, South Carolina
  - Clarksville, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Bellaire, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Irving, Texas
  - Nassau Bay, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Kirkland, Washington
  - Richland, Washington
  - Seattle, Washington
  - Clarksburg, West Virginia
  - Milwaukee, Wisconsin
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Mendoza
  - Santa Fe
- Chile (4):
  - Antofagasta
  - Arauco
  - Elqui
  - Santiago
- Colombia (4):
  - Bello, Antioquia
  - Antioquia
  - Barranquilla
  - Bogotá
- Mexico (6):
  - Mexicali, Estado de Baja California
  - León, Guanajuato
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Mérida, Yucatán
  - México

REFERENCES:
- [Derived] Mahableshwarkar AR, Calabrese JR, Macek TA, Budur K, Adefuye A, Dong X, Hanson E, Sachs GS. Efficacy and safety of sublingual ramelteon as an adjunctive therapy in the maintenance treatment of bipolar I disorder in adults: A phase 3, randomized controlled trial. J Affect Disord. 2017 Oct 15;221:275-282. doi: 10.1016/j.jad.2017.06.044. Epub 2017 Jun 20. PMID 28662460
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 100 investigative sites in Argentina, Chile, Colombia, Mexico and the United States from 21 December 2011 (first participants signed the informed consent form) to 26 March 2015.
Pre-assignment Details: Participants with a diagnosis of bipolar disorder were enrolled equally in 1 of 4 treatment groups, once a day placebo, Tak-375 SL (ramelteon) 0.1 mg, 0.4 mg or 0.8 mg.
Period: Overall Study
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Started | 164 | 164 | 160 | 154
Safety Analysis Set: Received Treatment | 163 | 164 | 159 | 154
Completed | 62 | 60 | 58 | 45
Not Completed | 102 | 104 | 102 | 109
Not completed — Pretreatment Event or Adverse Event | 9 | 4 | 6 | 5
Not completed — Major Protocol Deviation | 2 | 4 | 4 | 1
Not completed — Lost to Follow-up | 9 | 12 | 6 | 9
Not completed — Voluntary Withdrawal | 18 | 14 | 21 | 20
Not completed — Study Termination | 23 | 33 | 28 | 29
Not completed — Pregnancy | 0 | 1 | 1 | 3
Not completed — Relapse | 35 | 25 | 28 | 35
Not completed — Reason not Specified | 6 | 11 | 8 | 7

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg | Total
Number analyzed (Participants) | 164 | 164 | 160 | 154 | 642
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.21 (12.224) | 42.97 (13.262) | 42.93 (11.666) | 41.71 (12.534) | 42.98 (12.440)
Age, Customized [Number; unit: participants]
  <=50 Years | 109 | 105 | 113 | 112 | 439
  >50 Years | 55 | 59 | 47 | 42 | 203
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 89 | 92 | 90 | 367
  Male | 68 | 75 | 68 | 64 | 275
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 52 | 63 | 54 | 46 | 215
  Non-Hispanic and Non-Latino | 112 | 101 | 106 | 108 | 427
Race/Ethnicity, Customized [Number; unit: participants]
  White | 118 | 116 | 117 | 104 | 455
  Black | 36 | 34 | 34 | 36 | 140
  Asian | 1 | 1 | 1 | 4 | 7
  American Indian or Alaska Native | 5 | 8 | 5 | 4 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 1 | 3
  Multiple | 4 | 3 | 3 | 5 | 15
Region of Enrollment [Number; unit: participants]
  Argentina | 16 | 19 | 18 | 13 | 66
  Chile | 13 | 10 | 12 | 11 | 46
  Colombia | 4 | 7 | 7 | 6 | 24
  Mexico | 9 | 12 | 8 | 10 | 39
  United States | 122 | 116 | 115 | 114 | 467
Height [Mean (Standard Deviation); unit: cm] | 168.65 (10.159) | 168.56 (9.790) | 167.49 (10.235) | 168.47 (9.608) | 168.30 (9.943)
Weight [Mean (Standard Deviation); unit: kg] | 87.04 (21.148) | 87.52 (21.265) | 88.68 (22.291) | 85.71 (21.386) | 87.25 (21.500)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated using the weight collected at the first screening visit (Visit 1): BMI=weight(kg)/[height(m)]^2
  kg/m^2 | 30.68 (7.351) | 30.66 (6.382) | 31.52 (7.108) | 30.11 (6.702) | 30.75 (6.900)
Smoking Classification [Number; unit: participants]
  Participant Has Never Smoked | 75 | 69 | 75 | 62 | 281
  Participant is a Current Smoker | 56 | 68 | 58 | 63 | 245
  Participant is an Ex-smoker | 33 | 27 | 27 | 29 | 116
Participant Drinking Status [Number; unit: participants]
  Has Never Drunk | 68 | 70 | 65 | 58 | 261
  Ex-Drinker | 47 | 50 | 48 | 41 | 186
  Current Drinker | 49 | 43 | 47 | 55 | 194
  Missing | 0 | 1 | 0 | 0 | 1
If Drinker, Amount Consumed [Number; unit: participants] — Only participants with drinking status Current Drinker are accounted for: N=49, 43, 47, 55 in each treatment arm, respectively.
  participants
    <4 Drinks per Day | 49 | 42 | 47 | 55 | 193
    >= 4 Drinks per Day | 0 | 1 | 0 | 0 | 1
Does Participant Consume Caffeine? [Number; unit: participants]
  Yes | 121 | 122 | 122 | 127 | 492
  No | 43 | 42 | 38 | 27 | 150

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Any Relapse
Description: The time from randomization to relapse over 12 months double-blind treatment period as determined by the Principal Investigator (PI) or defined by any of the following criteria: depression [Montgomery-Åsberg Depression Rating Scale (MADRS) score ≥16]; mania/hypomania [Young Mania Rating Scale (YMRS) total score ≥14]; mixed episode [MADRS score ≥16 and YMRS total score ≥16]; or, whether participant receives psychiatric hospitalization for bipolar disorder, electroconvulsive therapy (ECT) or any psychotropic medication change prescribed for the treatment of depression, mania/hypomania or mixed episodes.
Time Frame: Randomization to Month 12 double-blind treatment period
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug and had at least one valid post-baseline value for assessment of primary efficacy. Participants without relapse were censored.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
Days | 248.3 (8.11) | 287.7 (8.83) | 253.1 (7.52) | 223.9 (7.60)
Statistical Analysis 1: Comparison: Placebo vs Ramelteon SL 0.1 mg; Test type: Superiority or Other; p = 0.286, Log Rank; Hazard Ratio (HR) = 0.77, 98.3% CI 2-sided [0.42 to 1.39] — Cox proportional hazards model with only treatment in the model
Statistical Analysis 2: Comparison: Placebo vs Ramelteon SL 0.4 mg; Test type: Superiority or Other; p = 0.332, Log Rank; Hazard Ratio (HR) = 0.78, 98.3% CI 2-sided [0.43 to 1.43] — Cox proportional hazards model with only treatment in the model
Statistical Analysis 3: Comparison: Placebo vs Ramelteon SL 0.8 mg; Test type: Superiority or Other; p = 0.808, Log Rank; Hazard Ratio (HR) = 1.06, 98.3% CI 2-sided [0.60 to 1.86] — Cox proportional hazards model with only treatment in the model
Statistical Analysis 4: Comparison: Placebo vs Ramelteon SL 0.1 mg; Test type: Superiority or Other; p = 0.286, Log Rank; Hazard Ratio (HR) = 0.88, 98.3% CI 2-sided [0.48 to 1.61] — Cox proportional hazards model with treatment, pooled center, age, gender, and baseline MADRS score in the model
Statistical Analysis 5: Comparison: Placebo vs Ramelteon SL 0.4 mg; Test type: Superiority or Other; p = 0.332, Log Rank; Hazard Ratio (HR) = 0.79, 98.3% CI 2-sided [0.42 to 1.49] — Cox proportional hazards model with treatment, pooled center, age, gender, and baseline MADRS score in the model
Statistical Analysis 6: Comparison: Placebo vs Ramelteon SL 0.8 mg; Test type: Superiority or Other; p = 0.808, Log Rank; Hazard Ratio (HR) = 1.08, 98.3% CI 2-sided [0.60 to 1.95] — Cox proportional hazards model with treatment, pooled center, age, gender, and baseline MADRS score in the model

2. Secondary Outcome: Time From Randomization to Relapse Due to Depression
Description: Relapse due to depression determined by any of the following criteria during the 12-month double-blind treatment period: PI judgment, MADRS ≥16, psychiatry hospitalization, ECT or any psychotropic medication change prescribed for the treatment of depressive episodes.
Time Frame: Randomization to Month 12 double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
Days | 256.5 (7.70) | 242.1 (5.56) | 260.8 (7.03) | 224.2 (6.31)

3. Secondary Outcome: Time From Randomization to Relapse Due to Mania/Hypomania or Mixed Episode
Description: Relapse due to mania/hypomania or mixed episode is determined by any of the following criteria: PI judgment, mania/hypomania [YMRS ≥16], mixed episode [MADRS ≥16 and YMRS ≥16], psychiatry hospitalization, ECT or any psychotropic medication change prescribed for the treatment of mania/hypomania or mixed episodes.
Time Frame: Randomization to Month 12 double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
days | 150.2 (1.60) | 319.3 (6.07) | 269.5 (3.69) | 255.5 (5.03)

4. Secondary Outcome: Time From Randomization to Relapse Due to Depression From PI Judgement and/or MADRS ≥16
Description: The time from randomization to relapse event during the 12 month double-blind treatment period due to depression, determined by the PI judgement and/or a MADRS score ≥16. MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60. Higher scores indicate greater severity of symptoms.
Time Frame: Randomization to Month 12 double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
days | 265.0 (7.14) | 245.1 (5.22) | 262.5 (6.90) | 224.2 (6.31)

5. Secondary Outcome: Time From Randomization to Relapse Due to Mania/Hypomania
Description: Relapse due to mania/hypomania is determined by the primary investigator (PI) judgement and/or a YMRS total score ≥16. YMRS is a 11 item scale with four items scale to assess manic symptoms, rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe), with 7 items rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe) with higher scores reflecting greater levels of mania. The YMRS total score is calculated as the sum of the 11 individual item scores and ranges from 0-60.
Time Frame: Randomization to 12 Month double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
days | 150.7 (1.60) | 328.8 (4.53) | 274.8 (2.20) | 263.3 (3.73)

6. Secondary Outcome: Time From Randomization to Relapse Due to Mixed Episode
Description: Relapse due to Mixed episode is determined by PI judgement and/or MADRS score ≥16 and YMRS total score ≥16. MADRS is a 10-item scale that measures overall severity of depressive symptoms rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60. YMRS is a four item scale to assess manic symptoms, rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe), with 7 items rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score is calculated as the sum of the 11 individual item scores and ranges from 0-60.
Time Frame: Randomization to Month 12 double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
days | 147.6 (0.63) | 150.2 (1.53) | 96.0 (0.89) | 180.5 (2.31)

7. Secondary Outcome: Time From Randomization to Relapse Due to Psychiatric Hospitalization for Bipolar Disorder
Description: The time from randomization to relapse event during the 12 months double-blind treatment period due to psychiatric hospitalization for bipolar disorder.
Time Frame: Randomization to Month 12 double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
days | 198.6 (2.29) | 34.8 (0.20) | 70.6 (0.52) | 251.3 (2.36)

8. Secondary Outcome: Time From Randomization to Relapse Due to Electroconvulsive Therapy (ECT) Administration
Description: The time from randomization to relapse event during the 12 month double-blind treatment period due to ECT.
Time Frame: Randomization to Month 12 double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
days | NA (NA) — No relapses due to ECT. | NA (NA) — No relapses due to ECT. | NA (NA) — No relapses due to ECT. | NA (NA) — No relapses due to ECT.

9. Secondary Outcome: Time From Randomization to Relapse Due to Psychotropic Medication Change Prescribed for the Treatment of Depression, Mania/Hypomania or Mixed Episodes
Description: The time from randomization to relapse event during the 12 month double-blind treatment period due to any psychotropic medication change prescribed for the treatment of depression, mania/hypomania or mixed episode(s).
Time Frame: Randomization to Month 12 double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
days | 197.8 (2.33) | 18.9 (0.13) | 257.9 (2.69) | 55.7 (0.46)

10. Secondary Outcome: Time From Randomization to Study Withdrawal for Any Reason
Description: The time from randomization to study withdrawal during the 12 month double-blind treatment period. Withdrawal includes pretreatment event/adverse event; liver function test abnormalities; major protocol deviation; lost to follow-up; voluntary withdrawal; study termination; pregnancy; lack of efficacy; participant has a depressive, mania/hypomania or mixed episode; is hospitalized for psychiatric reasons; receives electroconvulsive therapy for bipolar disorder; receives any psychotropic medication change prescribed for the treatment of depression, mania/hypomania or mixed episodes; or any other reason.
Time Frame: Randomization to Month 12 double-blind treatment period
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug and had at least one valid post-baseline value for assessment of primary efficacy.
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
days | 240.6 (11.44) | 226.8 (10.48) | 226.9 (10.88) | 208.7 (11.01)

11. Secondary Outcome: Quality of Life, Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) Total Score
Description: Q-LES-Q-SF is a self-administered 16-item questionnaire to assess the degree of enjoyment and satisfaction experienced by patients in various areas of daily functioning. It includes 30 items across five subscales (daily activities, clothing, diet/food habits, relationship, psychological well-being and distress), scored on a 6-point Likert scale with subscale and total score ranging from 0 (none) to 5 (all the time). For reporting purposes, the scores are reversed and higher scores reflect improved quality of life and positive changes relative to baseline indicate improved quality of life.
Time Frame: Baseline and Months 1, 2, 3, 4, 5, 6, 7, 8, 10 and 12
Population: Participants from the Full Analysis Set, all randomized participants who received at least 1 dose of study drug and had at least one valid post-baseline value for assessment of primary efficacy, with available data.
Measure: Mean (Standard Deviation); unit: percent of maximum total score
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Number analyzed (Participants) | 157 | 162 | 154 | 149
percent of maximum total score
  Baseline (n=115, 129, 121, 118) | 65.7 (17.00) | 65.1 (16.57) | 68.6 (15.71) | 65.8 (15.09)
  Month 1 (n=113, 127, 121, 118) | 68.3 (14.68) | 68.5 (15.48) | 70.2 (14.76) | 68.1 (14.65)
  Month 2 (n=115, 128, 121, 118) | 67.3 (16.24) | 68.7 (15.11) | 70.6 (15.07) | 67.4 (15.68)
  Month 3 (n=115, 129, 121, 118) | 66.5 (15.89) | 69.0 (14.83) | 70.0 (15.68) | 66.2 (16.74)
  Month 4 (n=115, 129, 121, 118) | 66.8 (17.18) | 68.9 (15.67) | 69.3 (15.11) | 66.9 (17.08)
  Month 5 (n=115, 129, 121, 118) | 67.2 (16.43) | 69.6 (16.86) | 69.6 (15.22) | 66.0 (16.72)
  Month 6 (n=115, 129, 121, 118) | 67.1 (17.37) | 68.4 (17.41) | 68.1 (16.09) | 67.2 (16.41)
  Month 7 (n=115, 129, 121, 118) | 67.0 (16.80) | 70.4 (15.98) | 69.7 (15.80) | 65.8 (17.61)
  Month 8 (n=115, 129, 121, 118) | 67.7 (16.63) | 71.0 (15.17) | 69.0 (17.24) | 66.8 (17.10)
  Month 10 (n=115, 129, 121, 118) | 67.9 (16.91) | 71.1 (16.57) | 70.2 (15.41) | 66.5 (17.62)
  Month 12 (n=115, 129, 121, 118) | 67.5 (17.69) | 70.9 (16.54) | 70.0 (15.97) | 66.8 (17.77)

ADVERSE EVENTS:
Time Frame: Approximately 30 days after the last dose of study drug (up to 12 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Ramelteon SL 0.1 mg | Ramelteon SL 0.4 mg | Ramelteon SL 0.8 mg
Serious Adverse Events (participants affected / at risk) | 10/163 | 14/164 | 6/159 | 8/154
Other Adverse Events (participants affected / at risk) | 55/163 | 47/164 | 49/159 | 50/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=163) | Ramelteon SL 0.1 mg (N=164) | Ramelteon SL 0.4 mg (N=159) | Ramelteon SL 0.8 mg (N=154)
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 1
Mania (Psychiatric disorders) | 1 | 1 | 1 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 2 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2 | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Victim of crime (Social circumstances) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=163) | Ramelteon SL 0.1 mg (N=164) | Ramelteon SL 0.4 mg (N=159) | Ramelteon SL 0.8 mg (N=154)
Diarrhoea (Gastrointestinal disorders) | 7 | 10 | 2 | 5
Influenza (Infections and infestations) | 3 | 6 | 8 | 5
Nasopharyngitis (Infections and infestations) | 11 | 6 | 10 | 13
Upper respiratory tract infection (Infections and infestations) | 11 | 7 | 9 | 6
Headache (Nervous system disorders) | 13 | 14 | 14 | 10
Depression (Psychiatric disorders) | 9 | 6 | 7 | 15
Insomnia (Psychiatric disorders) | 11 | 8 | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.